CLINICAL TRIAL: NCT05457413
Title: Impact of Bariatric Surgery Induced Weight Loss on Women Fertility: A Prospective Cohort Study
Brief Title: Impact of Bariatric Surgery on Women Fertility
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: MS 392/2022
Record Dates: First submitted 2022-07-05; First posted 2022-07-14 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-01

CONDITIONS: Fertility Issues
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sleeve gastrectomy: Sleeve gastrectomy for weight loss
  Interventions: Procedure: Sleeve gastrectomy

INTERVENTIONS:
Procedure: Sleeve gastrectomy — Bariatric surgery

SUMMARY:
Obesity is a multifactorial risk factor for subfertility, in relation to chronic hormonal change induced by adipose tissue. This prospective cohort study aims to evaluate the impact of bariatric surgery induced weight loss on women fertility.

DETAILED DESCRIPTION:
Females undergoing sleeve gastrectomy will be assessed for improvement of fertility indicators

ELIGIBILITY:
Inclusion Criteria:

* Age from 20-40 years.
* BMI >35 kg/m2

Exclusion Criteria:

* Women with medical endocrinal disorders as DM, thyroid, hyperprolactinaemia, etc.
* Women using any hormonal treatment or fertility drugs like oral contraceptive pills and/or metformin.
* Women have any surgical complication intra-operatively or post operatively.
* Women refused to participate in the study.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Obese females undergoing sleeve gastrectomy
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Antimullerian hormone level | 3 months
  Change in antimullerian hormone level

SECONDARY OUTCOMES:
Change in serum FSH level | 3 months
Change in serum LH level | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Maii Nawara, Study Director — Associate professor
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Cairo/القاهرة, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Anonymous participants data will be available with principal investigator and director for any inquiries
Time Frame: Will be availabe after publishing for 2 years
Access Criteria: Will be with corresponding author if required